CLINICAL TRIAL: NCT07288281
Title: "Duration of Preoperative Clear Fluids Fasting in Patients Undergoing Liver Transplant. A Prospective Observational Study: the "Timbarc-1" a Pilot Study"
Brief Title: "Duration of Preoperative Clear Fluids Fasting in Patients Undergoing Liver Transplant"
Acronym: Timbarc-1
Status: Recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: KB/67/2025
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-06

CONDITIONS: Preoperative Clear Fluid Fasting; Liver Transplant Recipient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- liver recipient: liver transplant recipient undergoing liver transplantation in University Clinical Center of Medical University of Warsaw

SUMMARY:
The goal of this prospective observational study is to report the duration of preoperative clear fluids fasting in patients undergoing liver transplant. It will also learn about the relationship between the duration of preoperative clear fluids fasting and changes in hemodynamic variables and metabolic profile at various anesthesia and transplant phases. The main questions it aims to answer are:

* How long liver recipient fast from clear fluids before liver transplant?
* Is there any relationship between the duration of preoperative clear fluids fasting and changes in blood pressure and hear rate after the induction of anesthesia?
* Is there any relationship between the duration of preoperative clear fluids fasting and blood glucose concentration, blood lactate concentration and acid base balance during anesthesia for liver transplant?

DETAILED DESCRIPTION:
Clear fluids include water, certain juices without pulp (like apple or grape), clear sodas, tea or coffee without milk or cream, clear broth, sports drinks, gelatin, and popsicles without fruit pulp or yogurt.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective liver transplant

Exclusion Criteria:

* patients unable to give detailed answer on clear fluid fasting due to severe hepatic encephalopathy or cognitive impairment
* lack of written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver diseases scheduled for elective liver transplant at University Clinical Centre of Medical University of Warsaw
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
clear fluids fasting | before the induction of anesthesia
  duration of preoperative clear fluids fasting in patients undergoing liver transplant

OTHER OUTCOMES:
preoperative clear fluids fasting and changes in hemodynamic variables and metabolic profile | after patient's coming to the operating room before induction of anesthesia till the end of the anhepatic phase of liver transplantation (just before the repercussion of liver graft)
  The correlation between the duration of preoperative clear fluid fasting and changes in heart rate, mean arterial pressure, blood glucose concentration, blood pH, blood lactate concentration and standard base excess after the induction of anesthesia till the end of the anhepatic phase of liver transplantation.

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinical Centre of Medical University of Warsaw, Warsaw, Warszawa, Poland

IPD SHARING:
Plan to Share IPD: No